CLINICAL TRIAL: NCT00155857
Title: National Taiwan University Hospital
Brief Title: The Genetic Study of Primary Angle-Closure Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9100209868
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-06

CONDITIONS: Glaucoma
Keywords: glaucoma, genetic
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The purpose of this study is to evaluate the possible candidate gene of Primary Angle-Closure Glaucoma.

DETAILED DESCRIPTION:
Glaucoma has long been recognised as a leading cause of blindness, and that the scale of the problem will only increase with future population growth and increasing life expectancy (1).

The epidemiological information available in 1993 in the World Health Organization's (WHO) global data bank on blindness was reviewed by Thylefors and Négrel (1). They developed a simple model estimating the number of glaucoma blind people in each World Bank region. Primary open angle glaucoma (POAG) was judged to be responsible for three million blind, primary angle closure glaucoma (PACG) for two million, and for congenital glaucoma the figure was 200 000, giving a total of 5.2 million blind. This represents 15% of global blindness. The number of people affected by glaucoma was estimated to be about 20 million.

In 1996, Quigley used 111 published reports of glaucoma prevalence to construct a statistical model of the number of people affected by glaucoma worldwide (2). Data were included only if the study design, methods, and reported results met certain specific criteria. The countries of the world were arranged in seven groups according to similarities in ethnicity and presumed characteristics of glaucoma. For each region, the available age specific prevalence of OAG and ACG were applied to population projections for the year 2000. It was estimated that 66.8 million people were affected by OAG and ACG, with nearly equal numbers of people affected by each disease. Few prevalence studies described secondary glaucoma separately, but an estimate of six million for secondary glaucoma was reached, making a total, without childhood glaucoma, of around 73 million affected. Of these, 6.7 million were thought to be blind (2).

There was reliable epidemiologic evidence to suggest that PACG is more common among Eskimos (3) and Chinese (4). As POAG was common in the western countries, there was a large population at risk in Asia (5). PACG among Asians was more frequently chronic and has few symptoms (6). Therefore, persons might not be motivated by symptoms to present to medical attention until significant visual damage has occurred in this region. A population-based study of screening techniques for PACG was performed in the township of Jin Shan in rural Taiwan (7). This joint US-Taiwanese project, published in 1996, identified a target population of 5441 people aged 40 years and older, of whom 562 were examined. A gonioscopic examination was carried out on all subjects. PACG was diagnosed in people with a "narrow" angle and either an IOP >18 mm Hg, an increase in IOP 8 mm Hg on dark prone provocation test, or a previous "acute" episode of angle closure with an iridectomy. The diagnosis did not depend on the presence of a visual field defect or structural optic neuropathy. There were 17 people diagnosed as suffering PACG (3.0%). Only 35% of cases gave a history of symptoms characteristic of "acute" angle closure. Two of these 17 people (12%) were blind in both eyes (7). As aforementioned, Taiwan has a high prevalence of PACG, which usually leads to blindness ultimately. There are many reported studies on genes of POAG and normal-tension glaucoma from Asia, including Japan (14,21,29), China (25), and Korea (24). However, studies about genetics of PACG were lacking. Hence, in this study, we use the model of genomewide microsatellite genotyping with method of linkage disequilibrium to study the possible candidate gene of PACG. Then, we will further sequence the cDNA forPAX6 to find out the possible mutation in the family with well-defined pedigree.

ELIGIBILITY:
Inclusion Criteria:

* An occludable angle was defined as one in which less than 90° circumference of the pigmented trabecular meshwork was visible. Persons in whom primary angle-closure was suspected (PACS) had an occludable angle and no other abnormality. Primary angle closure (PAC) was diagnosed in persons with a normal visual field and optic disc but having an occludable angle and evidence of angle dysfunction. Dysfunctional features included elevated IOP (>19 mm Hg) or a positive darkroom-prone provocation test, peripheral anterior synechiae, pigment smearing in superior drainage angle, sequelae of acute angle closure (iris whorling or glaukomflecken), or a clear history of symptomatic angle closure with evidence of a peripheral iridectomy. An IOP of 19 mm Hg was chosen by taking the mean +2 SDs from other data on Sino-Mongoloid people.

Primary angle-closure glaucoma was diagnosed in subjects with an occludable drainage angle and glaucomatous optic neuropathy with compatible visual morbidity. Optic neuropathy was defined as a CDR of 0.7 or more, or asymmetry of 0.2 or more. In early to moderate cases (CDR of 0.7 or 0.8 or asymmetry of 0.2), a reproducible visual field defect was required to confirm the diagnosis. In advanced cases (CDR >=0.9 or CDR asymmetry >0.3), perimetric evidence of visual loss was not an absolute requirement. Primary angle-closure glaucoma was diagnosed if the disc was not visible, but iris stromal atrophy and whorling were seen in conjunction with a visual acuity less than 20/400.

Exclusion Criteria:

* Individuals are excluded if there is known ocular disease or insult that could predispose to myopia, such as retinopathy of prematurity or early-age media opacification, or if they had a known genetic disease associated with myopia, such as Stickler or Marfan syndrome.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2003-07; Study Completion 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, MD, PHD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan